CLINICAL TRIAL: NCT00141804
Title: A Randomized Multicenter Study to Compare Tacrolimus and MMF With Tacrolimus and Rapamycin in Patients After Renal Transplantation
Brief Title: Efficacy and Safety of Sirolimus in Combination With Tacrolimus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Proverum GmbH (Unknown); KKS Netzwerk (Network); Fujisawa GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SirTac 01; contract number DE-02-RG-74
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-08

CONDITIONS: Kidney Transplantation
Keywords: renal transplantation; immunosuppression; prevention of acute rejection
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
To study the efficacy and safety of the administration of Tacrolimus in combination with Sirolimus for the prevention of acute rejection in patients after renal transplantation

DETAILED DESCRIPTION:
Basic randomized clinical trial (multicentre) in primary KTX to assess the safety and efficacy of a tac/rapa vs a tac/MMF regimen. Tac trough levels in accordance with current standards in both arms. Steroids to be used to individual centre protocol. Rapa trough levels will be adjusted to 5-10 ng/ml. Up to now only few data (primate and clinical) on tac/rap combinations available.

ELIGIBILITY:
Inclusion Criteria:

* first kidney transplantation
* re-transplantation
* non-related living donor transplantation
* patients > 18 years
* patients have given their written consent after being informed
* female patients in the age of parity must consent to an effective birth control and submit a negative pregnancy test

Exclusion Criteria:

* related living donation
* patients with known HIV-anamnesis
* patients who need systemically administered immunosuppression for another indication than the prophylaxis of kidney graft rejection
* patients with present malignant disease
* patients with clinically significant, uncontrolled infectional disease and/or severe diarrhea, vomiting or active gastric ulcer
* patients who haven taken part in a clinical study in the past 28 days and/or receive (received) medication which is not licensed by the responsible health authority
* other reasons which depend on the assessment of the physician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2002-01; Study Completion 2005-06

PRIMARY OUTCOMES:
- time to first biopsy proven acute rejection episode at month 12
- graft failure at month 12
- discontinuation of study medication at month 12

SECONDARY OUTCOMES:
- patient and graft survival at month 12
- incidence and severity of biopsy proven acute rejection episodes and incidence of steroid-resistant acute rejection episodes at month 12
- Renal function at month 12 (S-creatinine, Cockgroft-Gault clearance)
- incidence and severity of infections at month 12
- incidence of adverse events at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Heiner H. Wolters, Dr. med., Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany